CLINICAL TRIAL: NCT07044505
Title: Exploring the Molecular and Cellular Composition of Uterine Lavage Specimens Collected at the Time of Gynecologic Surgery.
Brief Title: Molecular and Cellular Profiling of Uterine Lavage Collected During Gynecologic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-77882
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Gynecologic Cancer; Gynecologic Disease; Gynecological Surgery; Uterine Cancer
MeSH Terms: conditions — Genital Diseases, Female; Uterine Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group (Experimental): Participants undergoing gynecologic surgery who agree to uterine lavage collection intraoperatively for molecular and cellular analysis.
  Interventions: Procedure: Uterine Lavage

INTERVENTIONS:
Procedure: Uterine Lavage — Saline is introduced into the uterine cavity and retrieved during surgery to collect cells and fluid for downstream molecular and cellular analyses.

SUMMARY:
This study is a designed as a to test the clinical and technical feasibility of using this novel uterine lavage collection catheter to collected UL samples from up to 50 individuals undergoing gynecologic surgery and to describe the cellular composition of these samples. In order to do this, it is a prospective consecutively-enrolled cohort of 50 participants, all of who will receive the intervention of uterine lavage collection.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing gynecologic surgery with Stanford Healthcare
* Intact uterus and cervix
* At least one intact fallopian tube and ovary (on the same side)
* Aged 18 years or older
* Ability to understand and the willingness to provide written informed consent.

Exclusion Criteria:

* Known endometrial or cervical cancer or endometrial or cervical intraepithelial neoplasia
* Status post bilateral salpingectomy or tubal ligation
* Lack of consenting capacity
* Positive preoperative pregnancy test
* Active uterine bleeding (i.e. menses, etc.)
* Intrauterine device in place
* Non-English speaking (requires interpretor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Characterization of cellular composition in uterine lavage fluid | At time of gynecologic surgery
  Quantification and classification of cell types obtained from uterine lavage specimens using cytology and/or flow cytometry.

SECONDARY OUTCOMES:
Molecular profiling of uterine lavage specimens | At time of surgery
  Analysis of RNA, DNA, or protein expression profiles in collected lavage fluid.
Detection of inflammatory biomarkers in uterine lavage | At time of surgery
  Measurement of cytokines or other markers associated with uterine immune status or pathology.

CONTACTS AND LOCATIONS:
Overall Officials: James Ford, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States